CLINICAL TRIAL: NCT04927182
Title: Impact of Moderate Exercise Training on Vitals and Peak VO2 in Different Age Categories of Adult in COVID-19.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REC/00877 Nayab Saleem
Record Dates: First submitted 2021-06-14; First posted 2021-06-15 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate Exercise Training (Age Group 1; Young adult 17 -30 years) (Experimental)
  Interventions: Other: Moderate Exercise Training (Age Group 1; Young adult 17 -30 years)
- Moderate Exercise Training (Age Group 2; 31 to 45 years) (Experimental)
  Interventions: Other: Moderate Exercise Training (Age Group 2; 31 to 45 years)
- Moderate Exercise Training (Age Group 3; Above 45 years) (Experimental)
  Interventions: Other: Moderate Exercise Training (Age Group 3; Above 45 years)

INTERVENTIONS:
Other: Moderate Exercise Training (Age Group 1; Young adult 17 -30 years) — Supervised Moderate exercise training will be given. This protocol consisted of 3 types of exercises. This includes walking/jogging/running for 23 minutes cycling for 23 minutes and stepping for 5 minutes. The protocol will be performed in 50 minutes sessions thrice a week.
  Arms: Moderate Exercise Training (Age Group 1; Young adult 17 -30 years)
Other: Moderate Exercise Training (Age Group 2; 31 to 45 years) — Supervised Moderate exercise training will be given. This protocol consisted of 3 types of exercises. This includes walking/jogging/running for 23 minutes cycling for 23 minutes and stepping for 5 minutes. The protocol will be performed in 50 minutes sessions thrice a week.
  Arms: Moderate Exercise Training (Age Group 2; 31 to 45 years)
Other: Moderate Exercise Training (Age Group 3; Above 45 years) — Supervised Moderate exercise training will be given. This protocol consisted of 3 types of exercises. This includes walking/jogging/running for 23 minutes cycling for 23 minutes and stepping for 5 minutes. The protocol will be performed in 50 minutes sessions thrice a week.
  Arms: Moderate Exercise Training (Age Group 3; Above 45 years)

SUMMARY:
* To determine the impact of moderate exercise training on vitals (BP, HR) in different age categories of adult in COVID-19.
* To determine the Impact of moderate exercise training on Peak VO2 in different age categories of adult in COVID-19
* To determine muscle discomfort due to physical training.

DETAILED DESCRIPTION:
As of 30th January 2020, the outbreak of the novel coronavirus disease, later called COVID-19, was declared a Public Health Emergency. Governments' immediate protective measurements aim to slow down the ongoing spread of the COVID-19 disease.

Coronavirus had infected people exponentially. It has a typical symptom of influenza which includes fever, cough, fatigue sore throat and additional symptoms like breathlessness and diarrhea. There was no specific treatment to cure it and no vaccination to prevent it from further progression. The solitary solution for prevent of this virus was isolation and no gathering, which has caused people to sit in their houses and wash hands.

Literature shows that a significant larger reduction in Blood Pressure was observed in participant performing aerobic exercise. A study shows comparison between African and Asian population with hypertension indicates that Asian participant reduced more BP as compared to African .

ELIGIBILITY:
Inclusion Criteria:

* Cognitively intact
* Age categories (Young adult 17 -30, Middle age adults 31 to 45, old Age Above 45)
* SBP>120 mm Hg or DBP>80 mm Hg, and who had no physical limitations that precluded exercise participation were recruited from the general population from Pakistan in COVID era.
* No Regular Exercise since MARCH 2020 (start of COVID era) 3 months at least.

Exclusion Criteria:

* Participant failing to fall in this category would be excluded of the study.
* Uncontrolled hypertension
* Major joint impairment
* Bone fracture in the last 6 months
* Asthmatic patients

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Modified Borg Scale of Perceived Exertion | 6th week
  Changes from the Baseline, It is a subjective numeric scale ranging from 0 to 10, where 0 indicates "no dyspnea" and 10 indicates "unbearable dyspnea." A number is chosen by the patient in order to decide the best score that matches his level of dyspnea during physical activity.
Systolic and diastolic blood pressure | 6th week
  Changes from the Baseline, Systolic Blood pressure (SBP) and Diastolic Blood Pressure (DBP) will be measured through sphygmomanometer
Nordic Musculoskeletal questionnaire | 6th Week
  The Nordic Musculoskeletal Questionnaire (NMQ) quantifies musculoskeletal pain and activity prevention in 9 body regions. The Nordic general questionnaire is a standardized instrument used to analyse musculoskeletal symptoms in an ergonomic or occupational health context. The NMQ is comprised of just 3 questions regarding musculoskeletal pain including annual and 7-day prevalence of symptoms and annual prevention from normal work (at home or away from home). For each Question body region wise; Yes and No options are there to report. Patient can report more than 1 body region.
6 Min walk test (Distance in meters) | 6th Week
  Changes from the baseline, 6 Min Walk Distance (6 MWD) was used to measure Functional capacity. It is a sub maximal exercise test which can aid in assessing functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters which an individual covers in 6 min without any support.
Peak VO2 with formula | 6th week
  A generalized equation can be used to determined peak VO2 (Peak rate of oxygen consumption). The generalized equation can be used to accurately estimate mean peak VO2 from mean 6 MWD, among groups of patients with diverse diseases without the need for cardiopulmonary exercise testing. The equation is:
  Mean peak VO2(ml/kg/mins) = 4.948 + 0.023*Mean 6 MWD (meter) Changes From the Baseline will be measured
Heart Rate/Pulse Rate | 6th week
  Changes from baseline, Pulse rate was measured per minute through pulse oximeter. Crossly it was measure by Chest belt (Polar HR monitors). Changes from the Baseline will be measure.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- General Population, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No